CLINICAL TRIAL: NCT00778739
Title: A Two-Way Crossover, Open-Label, Single-Dose, Fed, Bioequivalence Study of Cefprozil 250 mg/5 mL Oral Suspension Versus Cefzil TM Powder for Oral Suspension (250 mg/5 mL) in Normal Healthy Non-Smoking Male and Female Subjects
Brief Title: Bioequivalence Study of Cefprozil 250 mg/ 5mL Powder For Oral Suspension Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Laboratories
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 3079
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2008-10-23 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: bioequivalence 1) CEFPROZIL FOR ORAL SUSPENSION USP 250 mg/ 5 mL fed conditions
MeSH Terms: interventions — Cefprozil; Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): CEFPROZIL FOR ORAL SUSPENSION USP 250 mg/ 5 mL
  Interventions: Drug: CEFPROZIL FOR ORAL SUSPENSION USP 250 mg/ 5 mL
- 2 (Active Comparator): CEFPROZIL FOR ORAL SUSPENSION USP 250 mg/ 5 mL
  Interventions: Drug: CEFPROZIL FOR ORAL SUSPENSION USP 250 mg/ 5 mL

INTERVENTIONS:
Drug: CEFPROZIL FOR ORAL SUSPENSION USP 250 mg/ 5 mL

SUMMARY:
The study was conducted as an open-label, randomized, 2-way crossover study to compare the single-dose relative bioavailability of Cefprozil 250 mg/5 mL Oral suspension versus Cefzil TM Powder for Oral Suspension (250 mg/5 mL) following one 5 mL dose under fed conditions

DETAILED DESCRIPTION:
The study was designed to compare the rate and extent of absorption of cefprozil from the following products under fed condition:

1. CEFPROZIL FOR ORAL SUSPENSION USP 250 mg/ 5 mL (Ranbaxy Laboratories Limited, India)
2. Cefzil ® (CEFPROZIL) for oral suspension equivalent to 250mg/5mL anhydrous, cefprozil (Bristol-Myers Squibb Company USA) The bioequivalence of these formulations was assessed for cefprozil (Bristol-Myers Squibb Company, USA)

Thirty -two subjects (32) were recruited for the study of which 16 were males and 16 were females. All of them completed the study

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoking male or female with a minimum age of 18 years
2. Body Mass Index (BMI= weight/ height) greater than or equal to 18.5 kg/m3 and less than or equal to 29.9 kg/m3
3. Normal findings in physical examination, 12- lead ECG and vital signs (blood pressure between 100-140/60-90 mm Hg, heart rate between 50-90 beats/min, temperature between 35.8°C and 37.5 °C
4. Negative for drug abuse, nicotine, hepatitis B-surface antigen, hepatitis C and HIV, and for female subjects pregnancy serum (serum β-CG)
5. No clinical laboratory values outside of the acceptable range as defined by BCR, unless the Principal Investigator decided that they were not clinically significant
6. Female subjects who were surgically sterile for at least 6 months or post -menopausal for one year, or who avoided pregnancy prior to the study, during the study and up until one month after end of the study
7. Availability of the subject for the entire study period and willingness to adhere to the protocol requirements as evidenced by signed ICF

Exclusion Criteria:

Subject candidates who met the following criteria were excluded::

1. Known history of hypersensitivity to cefprozil (e.g. Cefzil TM , cephalosporin antibiotics or penicillin antibiotics
2. Known history or presence of cardiac, pulmonary, gastrointestinal, endocrine, musculoskeltal, neurological, hematological, liver or kidney disease, unless judged not clinically significant by the principal investigator or Sub-investigator.
3. Presence of any significant physical or organ abnormality
4. Any history or evidence of food allergies
5. Any subject with history of drug abuse
6. Any significant illness
7. History of colitis
8. Significant recent history of Asthma
9. Any history of severe allergic reaction
10. Any subject with recent hi story of alcohol abuse
11. Use of any prescription medication within 14 days preceding study
12. Use of OTC medication within 7 days before study
13. Female subjects: use of contraceptives (oral, transdermal, implant, Mirena ®) within 30 days prior to drug administration or a depot injection of progesterone drug (eg. Depo-Provera®) within one year prior to drug administration
14. Female subjects with evidence of pregnancy or lactation
15. Any subject with blood drawn prior to the study during the conduct of clinic study other than BCR or within lock out period specified by previous study conducted by BCR
16. Participation in clinical trial with investigational drug within 30 days preceding study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2005-06; Primary Completion 2005-06 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- Biovail Contract Research,, Toronto, Ontario, Canada

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html